CLINICAL TRIAL: NCT00004192
Title: A Randomized, Multicenter, Open-Label Study of Single Dose Filgrastim-SD/01 Versus Daily Filgrastim Following ESHAP Chemotherapy for Non-Hodgkin's Lymphoma
Brief Title: Colony-Stimulating Factors to Relieve Neutropenia in Patients With Recurrent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0272-99-FB; P30CA036727 (NIH); AMGEN-990117 (Other Grant/Funding Number: Amgen, Inc.); CWRU-AMGN-1499 (Other: Ireland Cancer Center); UCLA-9906080 (Other: Jonsson Comprehensive Cancer Center, UCLA); NCI-G99-1648 (Registry Identifier: National Cancer Institute)
Record Dates: First submitted 2000-01-21; First posted 2004-06-25 (Estimated); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma; Neutropenia
Keywords: neutropenia; Waldenstrom macroglobulinemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Neutropenia; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; pegfilgrastim; Cisplatin; Cytarabine; Etoposide; etoposide phosphate; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Intervention Model Description: This is a randomized, open label, multicenter study. Patients are randomized to one of two treatment arms. All patients receive etoposide IV over 1 hour on days 1-4, cisplatin IV continuously on days 1-4, methylprednisolone IV over 15 minutes on days 1-5, and cytarabine IV over 2 hours on day 5. Treatment is repeated every 21 days for up to 4 courses. Arm I: Patients receive filgrastim-SD/01 subcutaneously (SQ) on day 6. Arm II: Patients receive filgrastim (G-CSF) SQ daily beginning on day 6 and continuing for 12 days or until blood counts recover.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Dose Filgrastim (SD/01) (Experimental): Participants receive etoposide IV over 1 hour on days 1-4, cisplatin IV continuously on days 1-4, methylprednisolone IV over 15 minutes on days 1-5, and cytarabine IV over 2 hours on day 5. Treatment is repeated every 21 days for up to 4 courses. Arm I: Participants receive filgrastim-SD/01 subcutaneously (SQ) on day 6.
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cytarabine; Drug: etoposide; Drug: methylprednisolone
- Daily Filgrastim (G-CSF) (Experimental): Participants receive etoposide IV over 1 hour on days 1-4, cisplatin IV continuously on days 1-4, methylprednisolone IV over 15 minutes on days 1-5, and cytarabine IV over 2 hours on day 5. Treatment is repeated every 21 days for up to 4 courses. Arm II: Participants receive filgrastim (G-CSF) SQ daily beginning on day 6 and continuing for 12 days or until blood counts recover.
  Interventions: Biological: pegfilgrastim; Drug: cisplatin; Drug: cytarabine; Drug: etoposide; Drug: methylprednisolone

INTERVENTIONS:
Biological: filgrastim
  Other Names: Neupogen
  Arms: Single Dose Filgrastim (SD/01)
Biological: pegfilgrastim
  Other Names: Neulasta
  Arms: Daily Filgrastim (G-CSF)
Drug: cisplatin
  Other Names: chemotherapy drug
Drug: cytarabine
  Other Names: cytosine arabinoside
Drug: etoposide
  Other Names: Etopophos, Toposar
Drug: methylprednisolone
  Other Names: Depo-Medrol, Medrol, Solu-Medrol, P-Care D80, ReadySharp Methylprednisolone, and P-Care D40

SUMMARY:
RATIONALE: Colony-stimulating factors may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Randomized phase II trial to compare the effectiveness of filgrastim-SD/01 with that of filgrastim to relieve the neutropenia following combination chemotherapy in patients who have non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effect of single dose filgrastim-SD/01 vs daily filgrastim (G-CSF) on the duration of neutropenia in course 1 after combination chemotherapy in patients with recurrent non-Hodgkin's lymphoma. II. Compare the effect of these regimens on duration of neutropenia in courses 2-4, absolute neutrophil counts (ANC) in courses 1-4, time to ANC recovery in courses 1-4, and safety in these patients. III. Determine the pharmacokinetic profile of these drugs in course 1 in these patients.

OUTLINE: This is a randomized, open label, multicenter study. Patients are randomized to one of two treatment arms. All patients receive etoposide IV over 1 hour on days 1-4, cisplatin IV continuously on days 1-4, methylprednisolone IV over 15 minutes on days 1-5, and cytarabine IV over 2 hours on day 5. Treatment is repeated every 21 days for up to 4 courses. Arm I: Patients receive filgrastim-SD/01 subcutaneously (SQ) on day 6. Arm II: Patients receive filgrastim (G-CSF) SQ daily beginning on day 6 and continuing for 12 days or until blood counts recover.

PROJECTED ACCRUAL: A total of 60 patients (30 per arm) will be accrued for this study within at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-Hodgkin's lymphoma (NHL)

  o Relapsed disease or Refractory to first line cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) chemotherapy
* Age 18 and over
* ECOG 0-2Absolute neutrophil count at least 1,500/mm3Platelet count at least 150,000/mm3
* Creatinine not greater than 1.5 mg/dL or Creatinine clearance greater than 60 mL/min
* Fertile patients must use effective barrier contraception
* At least 4 weeks since prior radiotherapy
* At least 72 hours since prior antimicrobials
* At least 30 days since other prior investigational drug

Exclusion Criteria:

* No myelodysplastic syndrome or chronic myeloid leukemia
* Not pregnant or nursing/Negative pregnancy test
* No other prior malignancy except

  * Curatively treated basal cell or squamous cell carcinoma
  * Carcinoma in situ of the cervix
  * Surgically cured malignancy
* No hypersensitivity to E. coli derived products (e.g., filgrastim (G-CSF), insulin, asparaginase)
* No prior bone marrow or peripheral blood stem cell (PBSC) transplantation for NHL
* No prior filgrastim-SD/01
* No other concurrent myelopoietic growth factors
* No concurrent WBC transfusions
* No concurrent PBSC collection
* No more than 2 prior courses of chemotherapy for any malignancy
* No concurrent corticosteroids except topical steroids or as pre-medications or associated with chemotherapy
* No other concurrent investigational drug
* No concurrent prophylactic antibiotics during course 1

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2000-05-01 (Actual); Primary Completion 2001-02-01 (Actual); Study Completion 2001-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, Study Chair — University of Nebraska
Locations (3):
- United States (3):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Ireland Cancer Center, Cleveland, Ohio